CLINICAL TRIAL: NCT04584697
Title: A Randomized, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics and Efficacy of a Single Dose of STI-2020 (COVI-AMG™) in Outpatients With COVID-19 Who Are Asymptomatic or Have Mild Symptoms
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Efficacy of STI-2020 (COVI-AMG™) in Outpatients With COVID-19
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Different study will be conducted
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMG-COV-102
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020

STUDY DESIGN:
Intervention Model Description: Initially, 2 subjects will be enrolled at the 40 mg dose level. If no safety concerns arise, 48 subjects will then be randomized 1:1:1:1 to receive 40 mg COVI-AMG, 100 mg COVI-AMG, 200 mg COVI-AMG, or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- COVI-AMG (Experimental): A single injection of 40 mg, 100 mg, or 200 mg of COVI-AMG will be given on Study Day 1. Standard of care will be maintained for all subjects throughout the study.
  Interventions: Biological: COVI-AMG
- Placebo (Placebo Comparator): A single injection of placebo will be given on Study Day 1. Standard of care will be maintained for all subjects throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-AMG — COVI-AMG is a fully human SARS-CoV-2 neutralizing monoclonal antibody (mAb).
  Other Names: STI-2020
  Arms: COVI-AMG
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled study to assess the safety, PK profile, and efficacy of COVI-AMG in subjects with COVID-19.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study followed by an expansion cohort phase designed to investigate the safety, PK profile, and efficacy of a single injection of COVI-AMG in outpatient subjects with COVID-19 but are not likely to require hospital admission within 24 hours. Subjects will receive one of the following treatments: 40 mg COVI-AMG, 100 mg COVI-AMG, 200 mg COVI-AMG, or placebo. Subjects will be followed for 60 days after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Must be COVID-19 positive by RT-PCR or an equivalent test, using an appropriate sample such as nasopharyngeal [NP], nasal, oropharyngeal [OP], or salivary) ≤ 72 hours prior to randomization. A historical record of positive result from test conducted ≤ 72 hours prior to randomization is acceptable if it can be documented.
* Must be asymptomatic OR have mild symptoms but not requiring imminent (within 24h) hospitalization.
* Must be willing and able to comply with all planned study procedures and be available for all study visits and follow-up as required by this protocol.
* Subject or family member/caregiver must have provided written informed consent which includes signing the institutional review board approved consent form prior to participating in any study related activity.

Exclusion Criteria:

* Have a documented infection other than COVID-19 that requires systemic treatment or in the investigator's opinion could interfere with the participant's safety or interfere with the assessments if enrolled in the study.
* Have any medical condition that, in the Investigator's opinion, could adversely impact safety.
* Be pregnant or lactating and breast feeding
* Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, monoclonal antibodies (mAbs) against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit. Note: subjects who have been prescribed hydroxychloroquine or chloroquine with or without azithromycin or other approved products for the off-label treatment of COVID-19 prior to study enrollment may be included and may continue to receive these agents so long as the dose remains stable. Additionally, any approved or authorized treatment (e.g., remdesivir, dexamethasone or treatments approved under an Emergency Use Authorization) is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events by type, frequency, severity, and causality (safety) | Randomization through study completion at Day 60
  Safety as assessed by incidence of adverse events by type, frequency, severity, and causality
Incidence of treatment-emergent adverse events by type, frequency, severity, and causality (safety) | Randomization through study completion at Day 60
  Safety as assessed by incidence of treatment-emergent adverse events by type, frequency, severity, and causality
Incidence of serious adverse events by type, frequency, severity, and causality (safety) | Randomization through study completion at Day 60
  Safety as assessed by incidence of serious adverse events by type, frequency, severity, and causality
Incidence of dose-limiting toxicities (safety) | Randomization through study completion at Day 60
  Safety as assessed by incidence of dose-limiting toxicities
Incidence of clinically meaningful laboratory abnormalities (safety) | Randomization through study completion at Day 60
  Safety as assessed by incidence of clinically meaningful laboratory abnormalities
Viral load as assessed using plasma and salivary samples at various timepoints | Randomization through study completion at Day 60
  Viral load as assessed using plasma and salivary samples at various timepoints correlated with nasopharyngeal testing
Time from onset of COVID-19 symptoms to treatment (Day 1) | Day 1
  Time from onset of COVID-19 symptoms to treatment (Day 1)
Presence and levels of anti-drug antibodies directed to COVI-AMG | Randomization through study completion at Day 60
  Presence and levels of anti-drug antibodies directed to COVI-AMG
Cytokine levels post-treatment | Randomization through study completion at Day 60
  Cytokine levels post-treatment including EGF, IFNγ, IL-1β, IL-6, IL-8, IL-10, and TNFα will be measured by ELISA

SECONDARY OUTCOMES:
AUC of COVI-AMG (PK) | Randomization through study completion at Day 60
  Area under the serum concentration-time curve (AUC) of COVI-AMG
Cmax of COVI-AMG (PK) | Randomization through study completion at Day 60
  Maximum observed serum concentration (Cmax) of COVI-AMG
Tmax of COVI-AMG (PK) | Randomization through study completion at Day 60
  Time to Cmax (Tmax) of COVI-AMG
t½ of COVI-AMG (PK) | Randomization through study completion at Day 60
  Apparent serum terminal elimination half life (t½) of COVI-AMG

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343